CLINICAL TRIAL: NCT06909279
Title: The More Than Words® Program for Parents of Young Children With Social Communication Challenges: A Pilot Pragmatic Randomized Waitlist-Control Trial
Brief Title: Caregiver Training to Support Children With Social Communication Challenges
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Collaborators: The Hanen Centre, Toronto (Unknown)
Responsible Party: Principal Investigator, Janis Oram, Full Professor, Western University, Canada
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 126148
Record Dates: First submitted 2025-03-26; First posted 2025-04-03 (Actual); Last update posted 2025-05-11 (Actual); Status verified 2025-05

CONDITIONS: Autism Spectrum Disorder; Suspected Autism; Social Communication Challenges
Keywords: Autism; Parent mediated; Hanen More Than Words; Tele practice; Social communication challenges; pilot pragmatic RCT; virtual care
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder

STUDY DESIGN:
Intervention Model Description: This will be a pilot pragmatic, randomized waitlist controlled trial design, where participants will be randomly assigned to either the virtual MTW Treatment Group (TG) or a Waitlist Control Group (WCG). By focusing on real-world implementation, this will allow us to capture how the MTW program operates outside of controlled environments.
Who Masked: Outcomes Assessor
Masking Description: Because we are comparing receipt of a behavioural intervention to no treatment (waitlist for the treatment), masking of the participants and care providers is not possible. Outcome assessors conducting data entry and coding will be masked. Masking will be accomplished using de-identified participant ID numbers that do not identify group assignment and randomize the actual order in which repeated measures were collected .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Virtual MTW Treatment Group (TG) (Experimental): The TG will receive the MTW program which consists of (a) an orientation session, (b) a pre-program consultation appointment, (c) eight 2½ hour group training sessions (8-10 parents/group), and (d) three individual video feedback sessions. At the orientation session, the SLP provides an overview of the program, and provides the parent with two assessment forms to complete (i.e., parent report measures of their child's social communication and communicative participation). At the pre-program consultation, the SLP conducts an informal assessment of the child's communication and records a video of the parent-child interaction. Parents and SLPs co-develop communication goals based on the child's social communication needs and ability. During group training sessions, parents learn support strategies to target goals (e.g., joining a child's idea in play, rather than directing the play; using gestures and animated facial expressions to get the child's attention).
  Interventions: Behavioral: The Hanen Centre's More Than Words® program
- Waitlist Control Group (WCG) (No Intervention): The WCG will be in a waiting period for three months, after which they will receive the Hanen More Than Words® program. However, they can still access other services in their community to support their child during their waiting period.

INTERVENTIONS:
Behavioral: The Hanen Centre's More Than Words® program — The Hanen Centre's More Than Words® program is a globally used, parent coaching intervention delivered by speech-language pathologists (SLPs) to parents of children who have social communication challenges, which includes children with a confirmed or suspected diagnosis of autism. The training program is designed to provide parents with the tools, strategies, and support they need to help their children reach their full communication and social interaction potential.
  Arms: Virtual MTW Treatment Group (TG)

SUMMARY:
"More Than Words® - The Hanen Program® for Parents of Autistic Children or Children Who May Benefit from Social Communication Support" is a family-focused intervention program delivered by a speech-language pathologist (SLP). The goal of More Than Words is to empower parents to be the main facilitator of their child's social communication development, which increases the child's opportunities to develop social communication skills in everyday situations. It is one of the programs offered to families who receive services from Ontario's Preschool Speech and Language program, although some regions are not able to offer it at all or are only able to offer a shortened version of the program. The Hanen Centre recently made updates to the More Than Words program to allow it to be delivered virtually (online) and to align with the latest evidence.

Past research has found some evidence that the More Than Words program is effective, but knowledge is needed about the latest version of the program, including how effective it is when delivered online. It is important to understand who this program works best for and why. The purpose of the current study, called a pilot study, is to test a study plan that could be used in a future large study to answer these questions.

In this pilot study, the investigators will test procedures for comparing the outcomes of families who receive the More Than Words program to families who have not yet received it. Additionally, procedures for understanding varying responses to treatment will be tested. The study aims to determine whether the methods used for recruiting families, delivering the program, and monitoring progress are practical and function as expected in preparation for the future large-scale study.

DETAILED DESCRIPTION:
Background Pediatric speech-language pathologists (SLPs) report that a substantial proportion of their caseloads now include children with diagnosed or suspected autism. This aligns with persistent increases in autism diagnoses worldwide and underscores the importance of effective, feasible, and resource-efficient support services. For children with diagnosed autism, or children with social communication challenges who may be waiting for diagnostic assessments, identifying effective services targeting language and social communication is particularly important because development of these skills is among the most important contributors to long-term outcomes in autistic children. Furthermore, supporting social communication aligns with parents' treatment priorities for their autistic children.

SLPs provide early support services that focus on promoting engagement and communication within meaningful contexts. For young children, their parents are often their primary communication partners. Therefore, parent coaching interventions are commonly used by SLPs to support social communication development in young autistic children. Parent coaching interventions allow clinicians to capitalize on parents' expert knowledge of their child. These interventions increase the potential for children to generalize skills learned in sessions to their daily life, thus increasing treatment dosage without increasing the cost. Furthermore, by reducing the frequency of direct contact hours with the therapist, public systems can optimize resource use and make these interventions accessible to a greater number of parents.

The past decade has seen an increase in the number of randomized control trials (RCTs) examining the efficacy of parent-delivered early interventions for autistic children; however, most were conducted in specialized research clinics that often do not reflect how treatment is offered by community SLPs. This can negatively impact the generalizability of the findings to real-world clinical practice. While explanatory trials determine the efficacy of an intervention (in a highly controlled setting), pragmatic trials determine the effectiveness of an intervention in a real-world context, that is, everyday clinical practice. Pragmatic RCTs embrace the complexity, unpredictability, and inconsistency inherent in routine clinical practice by including diverse patient populations and allowing flexibility and variability in how the intervention is delivered. Additionally, few clinical trials have included examination of for whom the intervention works (moderators of treatment outcome), why the intervention works (mediators of treatment outcomes), or how implementation processes could have impacted treatment effects. This leaves clinicians with limited information to effectively individualize and refine interventions to fit child, family, and system needs.

One parent coaching intervention commonly used by SLPs is More Than Words® - The Hanen Program® for Parents of Autistic Children or Children Who May Benefit from Social Communication Support (MTW). In fact, a recent survey identified MTW as the preschool autism intervention program most widely used (61%) by SLPs in Ontario, Canada. The two existing RCTs on MTW involved university-based program delivery and report mixed findings that included positive effects in parents' responsiveness and aspects of social communication for some children. Non-randomized observational studies of the MTW program reported improved parent responsiveness, self-efficacy, and interaction style; and improved child language and social communication skills post-program. When asked about perceived outcomes, parents from community-delivered MTW programs highlighted the new strategies they learned, their child's growth in functional communication skills, overall improvement in their relationship with their child, and the social and professional support network they gained. Studies of parents' experiences participating in MTW suggests they value the program and the opportunity to connect with other parents, but seek improvements in navigating program content, the numerous forms associated with participation, parent-to-parent discussion, and the amount of individualized time with the SLP. Although these results are promising, as is the case for parent-delivered interventions more broadly, community-based RCTs of the MTW program are lacking, and little evidence exists for the mediators and moderators of effective MTW delivery in real-world practice. Pragmatic RCTs are needed to build this understanding.

For a pragmatic RCT of the MTW program (and other parent coaching interventions) to be useful, it is critical to ensure that the methods used to evaluate treatment effects and mediators/moderators are not only sound but also ecologically valid and feasible for use in the community practice contexts in which the study is to be conducted. Given that real-world practice can be highly variable and unpredictable in ways that are outside of the control of the researcher, large-scale RCTs can be at risk for implementation failure without careful attention at the methodological planning stages. One solution is to first conduct a pragmatic methodological feasibility trial to identify and develop mitigation plans for possible issues in recruitment, retention, data collection, and analysis. A second associated solution is to employ principles of integrated knowledge translation, that is, ensure that co-construction and collaboration between researchers and community partners begins right from the planning stages. This can ensure that outcome measures selected are ideal from both a reliability, validity, and sensitivity perspective and practical for clinicians and families to use during real-world program delivery. In sum, for a full-scale pragmatic RCT to be successful and for results to be meaningful to end users, foundational work is needed that focuses on (a) systematic co-development of a comprehensive evaluation protocol, (b) testing of the acceptability and feasibility of the evaluation protocol within real-world community settings, and subsequently, (c) pilot testing of a pragmatic RCT protocol.

Rationale With an overarching objective to conduct pragmatic RCTs of the MTW program, the investigators first needed a comprehensive evaluation protocol of the MTW program as implemented in community practice that would be both feasible for clinicians and families and sensitive enough to measure treatment effects and moderators and mediators of child and family outcomes. Therefore, the investigators partnered with program developers and expert SLPs from The Hanen Centre to co-construct a logic (causal) model of the MTW program that links specific program objectives with evaluation tools (outputs, outcomes) and procedures. In brief, key areas integrated during development of the logic model and evaluation plan included: (a) theories and research guiding MTW program development, (b) outcome measures and treatment mediators and moderators identified in previous research, (c) expert SLP views on MTW objectives and outcomes, and mediators and moderators affecting treatment responses, and (f) organizational structures, barriers, and facilitators for SLPs delivering the program. The result of this co-construction process was a logic model of the MTW program and an associated evaluation protocol with proposed outcome measures.

The investigators recently completed the second aim, which was to assess the feasibility of the selected outcome measures and proposed evaluation procedure ("A Single Arm Feasibility Study of a Caregiver-Delivered Intervention for Preschool-Aged Children with Social Communication Challenges"). The following dimensions of feasibility were assessed: (a) recruitment capability, (b) feasibility, acceptability, and practicality of data collection and analysis procedures, and (c) preliminary effectiveness based on the selected outcome measures. A pragmatic, single-arm, pre-post methodological feasibility study design was employed to implement our co-constructed evaluation protocol during MTW programs delivered by community-based SLPs as a part of standard care in the Ontario Preschool Language Program (PSL), a publicly-funded service. In brief, the results revealed that of those approached, 45% of SLPs and 57% of parent-child dyads were willing to participate. None of the 21 enrolled parent-child dyads withdrew from the study; however, outcome measure completion ranged from 48-81%, with 4 dyads providing little to no data. SLPs viewed study methods and measures as acceptable and feasible and researcher coding of video-recorded outcome measures was reliable and practical. Preliminarily effectiveness analyses showed post-program gains in children's early communication skills and communicative participation by parent report, and in 10 of 11 child, parent, and dyadic joint engagement behaviours coded by the researchers. All parents agreed or strongly agreed that their child benefited from the MTW program and most reported increased self-efficacy in supporting their child's communication.

Collectively, the results of the feasibility trial supported use of the investigators' co-constructed evaluation protocol in a future RCT of the MTW program. The current pilot RCT is the next step. The estimations of recruitment, retention, and adherence rates noted in the feasibility trial will provide valuable insights, allowing for observation of how new adjustments and procedures developed in response to these findings alter success in these components of the study procedures. This pilot RCT will also provide critical information on recruitment, retention, and data collection for the waitlist control group, which was not assessed in the previous study and for whom methodological uncertainties remain. Additionally, findings from the feasibility trial indicated that securing a sufficient number of community sites willing and able to randomize their patients was not feasible, as the program is already considered standard care despite limited definitive RCT data to support its use. Consequently, this pilot RCT has been designed to be as pragmatic as possible, aiming to simulate standard care while employing MTW program sessions specific to this study (i.e., sessions not already part of community SLPs' existing schedules).

Objectives The objective is to gather data that will inform the decision on whether to conduct, and refine the design of, a larger definitive RCT. This will be done by evaluating the feasibility of recruitment, randomization, retention, and adherence of parent-child dyads and exploring potential trends in the preliminary effectiveness of the virtual MTW program through a pilot pragmatic randomized waitlist control trial.

Methods The Virtual MTW Program in Ontario MTW is a 13-week parent-implemented program designed to enhance communication, play development, and parent-child interaction for children under 4 years of age who are autistic and/or have social communication challenges. MTW is delivered by SLPs certified by The Hanen Centre, a global not-for-profit organization based in Toronto that developed and routinely updates the program and trains SLPs in its delivery. Traditionally, MTW has been delivered in-person, but since the onset of the pandemic in 2020, a virtual version aimed at replicating the in-person experience was added. The program delivery model to be used in this study will be the virtual MTW program. Virtual delivery includes a group orientation session, a pre-program consultation appointment, eight 2½ hour group training sessions (typically with 6-8 parents per group), and three individual video feedback sessions. At the orientation session, the SLP provides an overview of the program and provides the parent with forms to complete (i.e., parent report of their child's communication, video consent form). At the pre-program consultation, the SLP conducts an informal assessment of the child's communication and records a video of the parent-child interaction. Parents and the SLP co-develop communication goals based on the child's social communication needs and ability. During group training sessions, parents learn support strategies to target goals (e.g., joining a child's idea in play, rather than directing the play). Group virtual education sessions include SLP-led didactic presentations, video examples, group discussions, and opportunities for practice (e.g., role play). During virtually delivered, individual video feedback sessions, parents demonstrate the use of communication facilitation strategies with their child, while the SLP records the interactions. The parent and SLP then review the videos together, analyze use of the strategies and how the child responded, and formulate plans to foster the development of new skills.

In Ontario, parents who have concerns about their young child's speech-language development can self-refer for services through the Ontario Preschool Speech and Language (PSL) program, a publicly funded provincial program supporting over 60,000 children from birth through to entry into senior kindergarten annually. For children with diagnosed or suspected autism in the Ontario PSL program, one common standard of care includes offering the MTW program to families. Some Ontario families elect to pursue privately funded SLP services instead. Although some private SLPs in Ontario may deliver the MTW group program as a part of their private services, this is less common.

For this pilot pragmatic RCT, registered SLPs employed by The Hanen Centre who routinely deliver MTW programs will deliver the program virtually according to their standard clinical delivery. For this study, recruitment of the parent-child participants and allocation to group program schedule will be independently conducted by the investigators

Participant Recruitment and Sample Size Recruitment will be complete through community SLPs across Ontario who provide services to children under 4 years. As such, most children will be recruited through their SLP in the Ontario PSL; however, SLPs in private practice who support this age range will also be sources of recruitment. The investigators will contact SLPs via email, directly for those in private practice or through regional managers for those working within the PSL program. A study flyer will be shared with SLPs for them to facilitate the recruitment of eligible parent-child dyads from their caseload for the study. Families will then self-refer if interested in participating.

Since pilot studies are not confirmatory trials and are hence not hypothesis driven, no formal sample size calculation will be carried out. Based on many literature studies, a sample size ranging from 12-35 is commonly recommended for conducting a pilot study. In the investigators' previous feasibility study, a recruitment rate of 57% was observed with 21 out of 37 parent-child dyads approached by SLPs enrolled in the study. There was no attrition; however, completion rates for pre-post outcome measures range from 60-70%. Based on these findings, the investigators aim to recruit 36 parent-child dyads for each of the two groups to target at minimum 15 complete datasets in each of the treatment and control groups.

Eligibility Pre-Screening. SLPs will share the study flyer with potential participants whom they believe to be eligible. Interested families will then be pre-screened for eligibility. Either they will complete an eligibility screening survey (delivered using REDCap, a secure, online data collection platform) by following the survey link from the flyer or they will contact the Study Coordinator by email/phone and answer pre-screening questions over the phone with the study coordinator or other study team member. As a part of this screening, parents are asked to confirm they are available to attend group sessions on either Saturday mornings or Monday evenings (or both).

Informed Consent. Families who screen eligible will be provided with a copy of the study consent form to download and review within the survey or will be sent a copy via email. A member of the research team will schedule a phone or Zoom call with the parent in which they will meet with a member of the research team to review the study information and consent form before e-signing it (in REDCap).

Measures Feasibility Outcome Measures. To examine the primary research questions related to the feasibility of the proposed RCT method, the following areas will be evaluated.

1. Recruitment. The number of participants who complete and pass the screening survey will be recorded. The number of participants who enroll (sign the consent form) will also be recorded.
2. Retention: To assess retention in the MTW program, parent's attendance over the duration of the program will be recorded by the Hanen SLP delivering the program. Study withdrawal and loss to follow-up will also be recorded.
3. Randomization: The randomization method will be assessed by comparing the treatment and waitlist control groups pre-program to ensure no significant difference between them in the baseline measures including child's age, sex, or CFCS Level.
4. Adherence: Completion rates for each baseline and treatment outcome measure at each time point will be recorded for both groups
5. Fidelity: A SLP fidelity measure was developed for this pilot RCT, to assess the Hanen SLP's ability to implement the program components as intended. The individual items in this measure represent content that SLPs delivering the program attend to, but do not necessarily explicitly document. As such, the self-administered, session-specific checklists in this measure aim to document what the SLP covers when delivering the group and individual sessions (in accordance with the MTW Program Leader's Guide that manualizes program delivery). After each session, the SLP indicates Yes (2), Partly (1), or No (0) about their ability to complete each program component associated with that session, which will be used to generate an overall session fidelity percentage score (total score/ total possible score x 100).

Demographic/Baseline Measures. These measures will be collected to describe sample characteristics, confirm group equivalence after randomization, and conduct exploratory mediator/moderator analyses.

1. Child and Family Questionnaire. This form was developed by the investigators to collect demographic information of the children and parents participating in this study. It includes details about the parent's relationship to the child, cultural and ethnic background, home language, education, and household income. For the child, it gathers information on age, sex assigned at birth, health conditions, developmental diagnoses, past or current interventions, and participation in an early learning environment. Additionally, it explores family history of speech, language, or learning difficulties.
2. Communication Function Classification System (CFCS). The CFCS is a valid and reliable tool used to classify a child's everyday communication abilities into one of five levels based on how they send and receive messages. The SLP assesses the child's current level of communication based on function not chronological age or developmental stage using the CFCS flow chart, which includes five levels ranging from Level I (Effective Sender and Receiver with unfamiliar and familiar partners) to V (Seldom Effective Sender and Receiver with familiar partners). As such, a lower level is indicative of greater effectiveness as a communicator.
3. MTW Social Communication Stage. The Social Communication Checklist is a Hanen Centre-developed MTW program form that is completed by SLPs in collaboration with parents. It is used to identify the stage that best describes the child's current communication skills according to stages addressed by MTW program and coined by The Hanen Centre as: Explorer, Requester, Early Communicator, and Partner. The number of checkmarks at each stage is tallied, with more checkmarks at higher stages indicative of better outcomes. The number of skills children gain at each stage from before to after the program will be counted.

Treatment Outcome Measures. A variety of child and parent treatment outcome measures will be recorded at baseline (T1 for TG; T1 and T2 for WCG), post-program (T2 for TG and T3 for WCG) and after 3 months of receiving the intervention (T3 for TG and T4 for WCG). These measures are described in the Outcome Measures section of the trial registration.

Following enrolment, the study coordinator will assign each parent-child dyad a unique study identification number, which will be linked to identifying information gathered through the consent process in a separate Master list.

Baseline Demographic Information Collection. Parents will receive an email with a link to Child and Family Questionnaire (a REDCap survey) to collect demographic and baseline information about the child, parent, and family. Additionally, an investigator who is (or is supervised by) a registered SLP will conduct the parent-child appointment remotely at a time convenient for parents. The purpose of this appointment is threefold: (a) to ask parents about their child's involvement in an early learning environment (a demographic data point for the Child and Family Questionnaire that requires discussion), (b) to discuss and observe the child's communication abilities in order to determine their current level of communication function, and (c) to review instructions for the parents to video record interactions with their child during the study. A semi-structured interview guide will be followed to ensure all three components are completed, and the research team member will code responses on a REDCap survey linked to the Child and Family Questionnaire previously completed by the parent.

Random Allocation. Once the above demographic/baseline information has been collected, parent-child dyads will be stratified according to their MTW group program availability (Saturdays and/or Mondays) in preparation for random allocation within these two strata. A maximum of 9 families can attend MTW program group sessions according to Hanen Centre requirements. As such, once 18 families enroll who are stratified into the same MTW group session day (Saturday or Monday), they will be randomly allocated to the TG (to receive the MTW intervention immediately) or the WCG (to receive the intervention after a 3-month waiting period). Given the relatively small sample size, blocked randomization stratified by session day availability will be employed. The randomization order will be generated in 3 blocks of 6 (3 TG and 3 WCG). To minimize the likelihood of more than three consecutive parent-child dyads being assigned to the same group, only 14 of the 20 possible block permutations will be used, with sequences TTWWWT, TWWWTT, WWWTTT, TTTWWW, WWTTTW, WTTTWW being eliminated. The study coordinator will use the following random sequence generator that follows these criteria for group allocation: https://www.online-python.com/GZQV5NHF6r. The same process will be repeated as each group of 18 families per stratum enroll. Depending on the rate and frequency of dyad recruitment, this means that overlapping Saturday and/or Monday MTW programs cohorts could occur during the study.

Once randomly assigned to groups, the study coordinator will contact families to inform them of their start dates, along with their scheduled time frames for completing study activities. A spreadsheet containing the names and contract information of the parent-child dyads for the TG will be provided to the Hanen SLP assigned to deliver that program session so that clinical contact and planning can begin. The same information for the WCG will be provided to the Hanen SLP assigned to that session ~3 weeks prior to its start date so as to minimize clinician awareness of families' allocation to TG versus WCG, recognizing that it may not be possible to fully mask order from the Hanen SLPs.

Outcome Measure Assessment Points. At each time point, parents will receive a reminder email that will include a link to the secure OneDrive folder specific to their family that will have a copy of two fillable PDF forms to be completed (FOCUS-34, CSBS-DP CQ) and instructions on how to record and upload their video interaction. Parents will collect 10-minute videotaped naturalistic interactions of themselves playing with their child and then upload them to their OneDrive folder. Included in the email will also be a link to the Parent and Services Evaluation (a REDCap survey), which includes questions about the past three months related to (a) parent's reported self-efficacy and (b) services and supports accessed for the child.

MTW Program. Once the family starts the MTW program, they will not be contacted by the investigators until after the program ends. During the pre-program consultation, the Hanen SLP will record the child's MTW social communication stage. Throughout the program, the Hanen SLP will record parent attendance and complete the corresponding SLP fidelity checklist to record their own fidelity to treatment for that session. These data will be uploaded by the Hanen SLP to a secure OneDrive folder unique to that SLP. The study coordinator will then abstract the social communication stage, adherence, and SLP fidelity into a case report form that uses only de-identified numbers for the dyads before submitting the data for analysis.

Video Coding. Following submission of all parent-child interaction videos, the video filenames will be de-identified by the study coordinator to mask both the group allocation and the time point of each video. Two trained and blinded research team members will code the JERI and Parent Fidelity from these video recordings, rating of each variable using REDCap forms. For all three measures, two coders will independently code 20% of videos to determine reliability using Cohen's Weighted Kappa.

Planned Analyses Analyses will primarily use descriptive statistics and confidence interval (CI) estimation to evaluate the study procedures and outcomes. Descriptive statistics will be used to characterize feasibility outcomes and participant measures at baseline and Times 1-4. Continuous variables (e.g., CSBS Total Raw Score, FOCUS-34) will be expressed as means and standard deviations (M ± SD), while categorical variables (e.g., JERI variables, CFCS levels, self-efficacy) will be presented as frequencies and percentages. Descriptive and statistical analyses will be conducted using JASP (Version 0.19.0).

A) Primary Feasibility Outcomes The summary below outlines the one overarching and five key progression criteria [hat will be evaluated using a traffic light system to determine whether a definitive RCT is feasible and what changes would be required (Green - RCT is feasible & no changes are needed, Amber - RCT is feasible following minor changes, Red - RCT is not feasible without major changes.) To assess baseline equivalences between the two groups, independent t-tests will be conducted in continuous measures and Fisher's exact test for categorical variables.

Objective 1: To evaluate overall feasibility of study procedures (recruitment, retention, randomization, data collection, data management, follow-up)

1. Green: Each component of the study procedures runs smoothly without serious problems or obstructions that were able to stop the study. Study procedures are judged strongly feasible and suitable to proceed by the study team and community collaborators.
2. Amber: Study procedures are judged to be likely feasible by the study team and community collaborators, but minor problems in one or more components of the study procedures need to be amended before proceeding
3. Red: The study team and community collaborators identified major problems in one or more components of the study procedures that must be remedied in order for the study to be feasible and to be able to proceed

Objective 2: To evaluate parent-child dyad recruitment rates

1. Green: 72 dyads are recruited (100%) within 9 months, with at least 30 dyads recruited within the first 4 months
2. Amber: 72 dyads are recruited but it takes longer than predicted (e.g.,12 months)
3. Red: Unable to recruit at least 36 (50%) dyads within 9 months

Objective 3: To evaluate parent-child dyad retention through to study completion

1. Green: ≥ 80% dyads retained to study completion (< 20% dropped out) in both the Treatment and Waitlist Control groups
2. Amber: 60-79% dyads retained to study completion in both the Treatment and Waitlist Control groups
3. Red: < 60% dyads retained to study completion in either the Treatment or the Waitlist Control group

Objective 4: To evaluate ability for randomization to yield baseline equivalence of groups

1. Green: Children in the Treatment and Control groups did not differ on baseline characteristics
2. Amber: Children in the Treatment and Control groups minimally differed in a few baseline characteristics
3. Red: Children in the Treatment and Control groups differed in multiple baseline characteristics

Objective 5: To evaluate adherence to outcome data completion.

1. Green: ≥ 80% completion rate (< 20% missing data) for all outcome measures at the pre- and post-treatment data collection points; and ≥ 70% completion rate for all measures at follow up
2. Amber: 60-79% completion rate for one or more outcome measures at the pre- and post-treatment data collection points; and/or 50-69% completion rate for one or more measures at follow up
3. Red: < 60% completion rate for one or more outcome measures at the pre- and post treatment data collection points; and/or < 50% completion rate for one or more measures at follow up

Objective 6. To evaluate SLP fidelity to treatment

1. Green: ≥80% of SLP sessions meet MTW fidelity standards (≥ 75% overall session fidelity percentage score)
2. Amber: 70-79% of SLP sessions meet MTW fidelity standards
3. Red: < 70% of SLP sessions meet MTW fidelity standards

(B) Secondary (Exploratory) Outcomes Although this study is not designed or powered to detect statistical effects, repeated measures ANOVA will be used to explore preliminary effectiveness, that is, possible changes within each group (TG and WCG) over time according to the treatment outcome measures. Post-hoc pairwise comparisons will explore differences between specific time points and groups. Given sample size limitations, p-values will not be examined. Effect sizes for time, group, and interaction effects will be calculated using Eta Squared (η²). The effect sizes will be reported, with thresholds interpreted as small (η² ≥ 0.01), medium (η² ≥ 0.06), and large (η² ≥ 0.14). 95% CIs will also be reported for the effect sizes. The Intention-To-Treat principle will be followed for these analyses.

Exploratory analyses aimed at identifying potential moderators and mediators of treatment effects will be conducted by combining data from the waitlist group after receiving the MTW program with the treatment group (maximum possible N=72). Potential moderators such child factors (e.g., age, functional communication level), parent factors (e.g., self-efficacy, level of education), and family context (e.g., household income, engagement in prior services, as well as mediators (e.g., parent self-efficacy, parent fidelity, early adoption of strategies) will be drawn from theoretically informed selection of variables including child factors and family context. Analyses will include visual inspection as well as examination of estimated effects, and 95% CIs.

ELIGIBILITY:
Inclusion criteria:

1. The child is under 48 months of age at the time of study enrolment.
2. The child has delays in social communication and play skills according to the clinical assessment of the child's community SLP.
3. The parent (or other primary caregiver) has a smart phone, tablet, or computer with webcam and internet access to attend the virtual MTW sessions and complete study measures
4. The parent is available to attend the 13-week virtual MTW program (which includes 9 online group sessions on Saturday mornings or Monday evenings).
5. The parent is comfortable communicating and filling out forms in English.

Exclusion Criteria:

Failure to meet the inclusion criteria outlined above.

Max Age: 47 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 72 (Estimated)
Dates: Start 2025-05-06 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Changes from baseline in Child Communicative Participation at post-program and follow-up | Within 2 weeks before the waitlist period (control group only), 2 weeks before program start, 2 weeks after program end, 13-15 weeks after program end
  The FOCUS-34 is a reliable and validated criterion-referenced measure of real-world changes in children's communicative participation in response to speech-language intervention. The FOCUS-34 includes 34 items based on the Activities and Participation components of the ICF. It includes 23 items focused on the child's capacity for communication and 11 items on the child's ability to engage independently, both of which parents rate on a 7-point Likert scale. The total score on the FOCUS-34 ranges from 34-238 points, although the primary clinical outcome is the pre-post-program change scores. A change score of 11 points or more is considered a meaningful clinical change, 7-10 is possibly a meaningful clinical change, and 6 or less is not likely a meaningful clinical change. The FOCUS-34 is used in the Ontario PSL as a provincial outcome monitoring tool and thus is part of the existing standard of care for participants in this study.
Changes from baseline in global social communication challenges at post-program and follow-up | Within 2 weeks before the waitlist period (control group only), 2 weeks before program start, 2 weeks after program end, 13-15 weeks after program end
  The Clinical Global Impression (CGI) is a tool designed to quickly and sensitively monitor patient progress within clinical trials and has been adopted for the purpose of evaluating social communication behaviors following delivery of brief clinical interventions. The CGI-Severity will be coded at each timepoint in response to the prompt, "How impacted is the participant by social communication challenges at this time?" using a 7-point severity scale (1-normal, 2-borderline, and 3-mildly, 4-moderately, 5-markedly, 6-severely, 7-extremely impacted). Post-program, CGS-Improvement will be coded to assess changes in social communication challenges relative to pre-program on a 7-point scale (1-very much improved, 2-much improved, 3-minimally improved, 4-no change, 5-minimally worse, 6-much worse, 7-very much worse), with higher Improvement ratings meaning worse outcomes.
Changes from baseline in joint engagement at post-program and follow-up | Within 2 weeks before the waitlist period (control group only), 2 weeks before program start, 2 weeks after program end, 13-15 weeks after program end
  The Joint Engagement Rating Inventory (JERI) is an observational measure designed to capture various features of joint engagement that occur between young children and their parents. The 2020 version of the JERI has 32 items, but as recommended in the manual, the investigators will use a subset of social engagement behaviors aligned with the specific research questions, namely, 11 items aligned with skills targeted by the MTW program. This includes five child behavioural outcomes (initiation of communication, responsiveness to partner's communication, expressive language level and use, quality of behaviour patterns, affect), four parent behavioural outcomes (affect, following in on the child's focus, symbol highlighting, scaffolding) and two dyadic interaction items (fluency and connectedness, routines and rituals). Each behavior item is scored on a 7-point rating scale (ranging from being 1-minimally to 7-highly present, with higher scores meaning better outcomes).
Changes from baseline in parent evaluation of self-efficacy and services at post-program and follow-up | Within 2 weeks before the waitlist period (control group only), 2 weeks before program start, 2 weeks after program end, 13-15 weeks after program end
  The Parent Self-Efficacy and Services Evaluation survey incorporates two self-efficacy questions from the Early Intervention Parenting Self-Efficacy Scale: (a) "I feel confident that I can help my child to communicate their thoughts and ideas" and (b) "I feel confident that I can help my child develop their play skills". Each question will be rated on a 7-point Likert scale (from 1-strongly agree to 7-strongly disagree, with higher scores meaning a worse outcome). The remaining questions ask parents to report on and evaluate the perceived effectiveness of any services or developmental supported received over the last 3 months (including the MTW program after they receive it).
Changes from baseline in child prelinguistic skills at post-program and follow-up | Within 2 weeks before the waitlist period (control group only), 2 weeks before program start, 2 weeks after program end, 13-15 weeks after program end
  The Communication and Symbolic Behavior Scales - Developmental Profile Caregiver Questionnaire (CSBS-DP CQ) contains 41 multiple-choice items that assess seven prelinguistic skills: emotion and eye gaze, communication (rate and communicative function), gestures, sounds, words, understanding, and object use (symbolic and constructive play). Three composite scores (social, speech, symbolic) and a total raw score are generated. Although designed for children aged 6 to 24 months, it can be used with older children who are functioning within this developmental range and thus is applicable to the target population of the MTW program. The investigators will record Social, Expressive Speech and Symbolic Communication composites and Total raw scores.
Changes from baseline in parent use of More Than Words strategies at post-program and follow-up | Within 2 weeks before the waitlist period (control group only), 2 weeks before program start, 2 weeks after program end, 13-15 weeks after program end
  The Parent Fidelity Scale was developed for this pilot RCT to assess parent's use of the MTW program communication facilitation strategies during interactions with their child. The scale includes 13 items reflecting the core strategies that are taught across the MTW program group sessions and that the SLP supports the parent to develop during the individual video feedback sessions. Each item will be rated on a 5-point Likert scale ranging from 1- Never/Rarely Used (never or only occasionally used the strategy, but almost all opportunities were missed) to 5 - Full Mastery (used the strategy effectively throughout the session, with very few or no missed opportunities). The rating scale will be coded from the same video-recorded interactions used for the JERI and CGI.

CONTACTS AND LOCATIONS:
Locations (1):
- Western University, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Given the sensitive nature of the research, data will not be available for sharing.

REFERENCES:
- [Background] Teare MD, Dimairo M, Shephard N, Hayman A, Whitehead A, Walters SJ. Sample size requirements to estimate key design parameters from external pilot randomised controlled trials: a simulation study. Trials. 2014 Jul 3;15:264. doi: 10.1186/1745-6215-15-264. PMID 24993581
- [Background] Julious SA. Sample size of 12 per group rule of thumb for a pilot study. Pharm Stati 2005;4:287-91
- [Background] Kunselman AR. A brief overview of pilot studies and their sample size justification. Fertil Steril. 2024 Jun;121(6):899-901. doi: 10.1016/j.fertnstert.2024.01.040. Epub 2024 Feb 6. PMID 38331310
- [Background] Gadke DL, Kratochwill TR, Gettinger M. Incorporating feasibility protocols in intervention research. J Sch Psychol. 2021 Feb;84:1-18. doi: 10.1016/j.jsp.2020.11.004. Epub 2020 Dec 4. PMID 33581765
- [Background] Binns, AV, Tucker P, Denusik L, Kumar, VR., & Oram J. The More Than Words® parent-delivered program for autistic children and those with social communication challenges: A single arm pragmatic feasibility trial. Pilot Feasibil Stud. Under review; 2025
- [Background] Binns AV, Kumar VR, Tucker T, Oram J. Co-constructing a logic model of the More Than Words program for real-world outcome evaluation. Unpublished manuscript. 2025.
- [Background] W.K. Kellogg Foundation. Using logic models to bring together planning evaluation and action: logic model development guide. Battle Creek, Michigan, USA: W.K. Kellogg Foundation; 2004. Available online: https://wkkf.issuelab.org/resource/logic-model-development-guide.html
- [Background] Patterson SY, Smith V. The experience of parents of toddlers diagnosed with autism spectrum disorder in the more than words parent education program. Infants Young Child. 2011;24(4):329-343. https://doi.org/10.1097/IYC.0b013e318229ebfd
- [Background] Denusik L, Servais M, Glista D, Hatherly K, Moodie S, Cardy JO, Weitzman E, Cunningham BJ. Families' Experiences in the Virtual Hanen More Than Words Program During the COVID-19 Pandemic. Am J Speech Lang Pathol. 2023 Mar 9;32(2):701-716. doi: 10.1044/2022_AJSLP-22-00256. Epub 2023 Mar 6. PMID 36877765
- [Background] Denusik L, Glista D, Servais M, Friesen J, Oram J, Cunningham BJ. "We were the best people to do the job": Caregivers' reported outcomes of a virtual caregiver-delivered program for autistic preschoolers. Autism Dev Lang Impair. 2024 Apr 30;9:23969415241244767. doi: 10.1177/23969415241244767. eCollection 2024 Jan-Dec. PMID 38694817
- [Background] Noyan Erbas A, Ozcebe E, Cak Esen T. Investigation of the effect of Hanen's "More Than Words" on parental self-efficacy, emotional states, perceived social support, and on communication skills of children with ASD. Logoped Phoniatr Vocol. 2021 Apr;46(1):17-27. doi: 10.1080/14015439.2020.1717601. Epub 2020 Jan 31. PMID 32003252
- [Background] McConachie H, Randle V, Hammal D, Le Couteur A. A controlled trial of a training course for parents of children with suspected autism spectrum disorder. J Pediatr. 2005 Sep;147(3):335-40. doi: 10.1016/j.jpeds.2005.03.056. PMID 16182672
- [Background] Girolametto L, Sussman F, Weitzman E. Using case study methods to investigate the effects of interactive intervention for children with autism spectrum disorders. J Commun Disord. 2007 Nov-Dec;40(6):470-92. doi: 10.1016/j.jcomdis.2006.11.001. Epub 2006 Dec 12. PMID 17169368
- [Background] Venker CE, McDuffie A, Ellis Weismer S, Abbeduto L. Increasing verbal responsiveness in parents of children with autism:a pilot study. Autism. 2012 Nov;16(6):568-85. doi: 10.1177/1362361311413396. Epub 2011 Aug 16. PMID 21846665
- [Background] Carter AS, Messinger DS, Stone WL, Celimli S, Nahmias AS, Yoder P. A randomized controlled trial of Hanen's 'More Than Words' in toddlers with early autism symptoms. J Child Psychol Psychiatry. 2011 Jul;52(7):741-52. doi: 10.1111/j.1469-7610.2011.02395.x. Epub 2011 Mar 22. PMID 21418212
- [Background] Sussman F, Drake L, Lowry L, Honeyman S. More than words: The Hanen program for parents of children with autism spectrum disorder or social communication difficulties. Hanen Centre Publication; 2016.
- [Background] Chan CL, Taljaard M, Lancaster GA, Brehaut JC, Eldridge SM. Pilot and feasibility studies for pragmatic trials have unique considerations and areas of uncertainty. J Clin Epidemiol. 2021 Oct;138:102-114. doi: 10.1016/j.jclinepi.2021.06.029. Epub 2021 Jul 3. PMID 34229091
- [Background] Binns AV, Smyth R, Andres A, Lam J, Oram Cardy J. Looking back and moving forward: A scoping review of research on preschool autism interventions in the field of speech-language pathology. Autism Dev Lang Impair. 2021 Oct 20;6:23969415211033171. doi: 10.1177/23969415211033171. eCollection 2021 Jan-Dec. PMID 36381535
- [Background] Iemmi V, Knapp M, Ragan I. Autism Dividend. Michael Smith Foundation for Health Research (MSFHR). 2017.
- [Background] Binns AV, Oram Cardy J. Developmental social pragmatic interventions for preschoolers with autism spectrum disorder: A systematic review. Autism Dev Lang Impairments. 2019;4. https://doi.org/10.1177/2396941518824497
- [Background] Volden J, Duku E, Shepherd C, Ba, Georgiades S, Bennett T, Di Rezze B, Szatmari P, Bryson S, Fombonne E, Mirenda P, Roberts W, Smith IM, Vaillancourt T, Waddell C, Zwaigenbaum L, Elsabbagh M; Pathways in ASD Study Team. Service utilization in a sample of preschool children with autism spectrum disorder: A Canadian snapshot. Paediatr Child Health. 2015 Nov-Dec;20(8):e43-7. doi: 10.1093/pch/20.8.e43. PMID 26744563
- [Background] Pituch K, Green V, Didden R, Lang R, O'Reilly M, Lancioni G, Sigafoos J. Parent-reported treatment priorities for children with autism spectrum disorders. Res Autism Spectr Disord. 2011;5:135-143. https://doi.org/10.1016/j.rasd.2010.03.003
- [Background] Denne LD, Hastings RP, Hughes CJ. Common approaches to intervention for the support and education of children with autism in the UK: an internet-based parent survey. Int J Dev Disabil. 2017 Jan 9;64(2):105-112. doi: 10.1080/20473869.2016.1275439. PMID 34141297
- [Background] Tidmarsh L, Volkmar FR. Diagnosis and epidemiology of autism spectrum disorders. Can J Psychiatry. 2003 Sep;48(8):517-25. doi: 10.1177/070674370304800803. PMID 14574827
- [Background] Baio J, Wiggins L, Christensen DL, Maenner MJ, Daniels J, Warren Z, Kurzius-Spencer M, Zahorodny W, Robinson Rosenberg C, White T, Durkin MS, Imm P, Nikolaou L, Yeargin-Allsopp M, Lee LC, Harrington R, Lopez M, Fitzgerald RT, Hewitt A, Pettygrove S, Constantino JN, Vehorn A, Shenouda J, Hall-Lande J, Van Naarden Braun K, Dowling NF. Prevalence of Autism Spectrum Disorder Among Children Aged 8 Years - Autism and Developmental Disabilities Monitoring Network, 11 Sites, United States, 2014. MMWR Surveill Summ. 2018 Apr 27;67(6):1-23. doi: 10.15585/mmwr.ss6706a1. PMID 29701730
- [Background] Binns AV, Cunningham BJ, Andres A, Oram Cardy J. Current practices, supports, and challenges in speech-language pathology service provision for autistic preschoolers. Autism Dev Lang Impair. 2022 Aug 29;7:23969415221120768. doi: 10.1177/23969415221120768. eCollection 2022 Jan-Dec. PMID 36382071